CLINICAL TRIAL: NCT00785733
Title: SMART Way of Treating Asthma. Non-interventional Study to Evaluate Clinical Efficacy of Symbicort® Maintenance And Reliever Therapy (Symbicort® SMART) in the Treatment of Patients With Moderate and Severe Asthma
Brief Title: NIS-observe Treatment Efficacy in Maintaining Symptoms Control in Moderate/Severe Asthma With Symbicort SMART
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Cristina Pentiuc, Medical Science Director, AstraZeneca
Other Study IDs: NIS-RRO-SYM-2008/1
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Moderate/Severe Asthma
Keywords: asthma
MeSH Terms: conditions — Lymphoma, Follicular; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Moderate and severe asthma patients stabilized on Symbicort SMART

SUMMARY:
The primary objective of this non-interventional study is to evaluate efficacy of Symbicort® SMART treatment in adult patients with moderate to severe asthma using ACQ scores during 6 months period

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for entry into study are the patients diagnosed with moderate to severe asthma, that the doctors have already decided to treat with Symbicort SMART within the last month, before inclusion in this program
* All eligible patients will be included in the protocol provided they will receive detailed information in advance and will sign consent to grant access to their own data collected during this programme.

Exclusion Criteria:

* All the patients who have a known hypersensitivity to Symbicort or any of its excipients will not be included in this study.
* As per valid Romanian SmPC, concomitant medication, that could result in drug interactions and could jeopardise patient safety will be carefully considered before having the patient enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The programme will include patients with moderate and severe asthma stabilized on Symbicort SMART from community sample
Sampling Method: Probability Sample
Enrollment: 1182 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire ACQ | 5 visits (V1-week 0, V2-week 4, V3-week 8, V4-week 16, V5-week 24)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Pentiuc, Study Chair — AstraZeneca
Locations (44):
- Romania (44):
  - Research Site, Alba Iulia
  - Research Site, Alexandria
  - Research Site, Arad
  - Research Site, Bacau
  - Research Site, Baia Mare
  - Research Site, Botoșani
  - Research Site, Brasov
  - Research Site, Brăila
  - Research Site, Breaza
  - Research Site, Bucharest
  - Research Site, Buftea
  - Research Site, Campulung Muscel
  - Research Site, Câmpina
  - Research Site, Călăraşi
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Deva
  - Research Site, Drobeta-Turnu Severin
  - Research Site, Giurgiu
  - Research Site, Hunedoara
  - Research Site, Iași
  - Research Site, Leordeni
  - Research Site, Miercurea-Ciuc
  - Research Site, Mizil
  - Research Site, Oradea
  - Research Site, Palazu Mare
  - Research Site, Piatra Neamţ
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Reşiţa
  - Research Site, Rm. Valcea
  - Research Site, Scorniceşti
  - Research Site, Sf. Gheorghe
  - Research Site, Sibiu
  - Research Site, Slobozia
  - Research Site, Suceava
  - Research Site, Târgovişte
  - Research Site, Târgu Mureş
  - Research Site, Tg. Jiu
  - Research Site, Timișoara
  - Research Site, Tulcea
  - Research Site, Vaslui
  - Research Site, Zalău